CLINICAL TRIAL: NCT02780141
Title: A Phase 3, Multi-center, Randomized, 2-arm, Open-label Study of Intermittent Oral Dosing of ASP1517 in Erythropoiesis Stimulating Agent-naive Hemodialysis Chronic Kidney Disease Patients With Anemia
Brief Title: A Study of Intermittent Oral Dosing of ASP1517 in Erythropoieses Stimulating Agent (ESA)-Naive Hemodialysis Chronic Kidney Disease Patients With Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1517-CL-0308
Record Dates: First submitted 2016-05-19; First posted 2016-05-23 (Estimated); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: ESA-naive Hemodialysis Chronic Kidney Disease Patients With Anemia
Keywords: Renal anemia; Roxadustat; ASP1517; Hemodialysis
MeSH Terms: interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASP1517 Low dose Group (Experimental): Study drug will be dosed three times weekly and dose adjustments will be made during the study.
  Interventions: Drug: roxadustat
- ASP1517 High dose Group (Experimental): Study drug will be dosed three times weekly and dose adjustments will be made during the study.
  Interventions: Drug: roxadustat

INTERVENTIONS:
Drug: roxadustat — Oral
  Other Names: ASP1517

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of ASP1517 in ESA-naive hemodialysis chronic kidney disease patients with anemia.

ELIGIBILITY:
Inclusion Criteria:

* Mean of the subjects' two most recent Hb values during the Screening Period must be ≤10.0 g/dL with an absolute difference ≤1.0 g/dL between the two values
* Either transferrin saturation (TSAT) ≥ 5% or serum ferritin ≥ 30 ng/mL during the screening period
* Female subject must either:

Be of non-childbearing potential:

* post-menopausal (defined as at least 1 year without any menses) prior to Screening, or
* documented surgically sterile Or, if of childbearing potential,
* Agree not to try to become pregnant during the study and for 28 days after the final study drug administration
* And have a negative pregnancy test at Screening
* And, if heterosexually active, agree to consistently use two forms of highly effective form of birth control (at least one of which must be a barrier method) starting at Screening and throughout the study period and continued for 28 days after the final study drug administration.

  * Female subject must agree not to breastfeed starting at Screening and throughout the study period, and continued for 28 days after the final study drug administration.
  * Female subject must not donate ova starting at Screening and throughout the study period, and continued for 28 days after the final study drug administration.
  * Male subject and their female spouse/partners who are of childbearing potential must be using two forms of highly effective form of birth control (at least one of which must be a barrier method) starting at Screening and continue throughout the study period, and for 12 weeks after the final study drug administration
  * Male subject must not donate sperm starting at Screening and throughout the study period and, for 12 weeks after the final study drug administration

Exclusion Criteria:

* Concurrent retinal neovascular lesion requiring treatment and macular edema requiring treatment
* Concurrent autoimmune disease with inflammation that could impact erythropoiesis
* History of gastric/intestinal resection considered influential on the absorption of drugs in the gastrointestinal tract (excluding resection of gastric or colon polyps) or concurrent gastroparesis
* Uncontrolled hypertension
* Concurrent congestive heart failure (NYHA Class III or higher)
* History of hospitalization for treatment of stroke, myocardial infarction, or pulmonary embolism within 12 weeks before the screening assessment
* Positive for hepatitis B surface antigen (HBsAg) or anti-hepatitis C virus (HCV) antibody at the screening assessment, or positive for human immunodeficiency virus (HIV) in a past test
* Concurrent other form of anemia than renal anemia
* Having received treatment with protein anabolic hormone, testosterone enanthate, or mepitiostane within 6 weeks before the screening assessment
* Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), or total bilirubin that is greater than the criteria, or previous or concurrent another serious liver disease at screening assessment
* Previous or current malignant tumor (no recurrence for at least 5 years is eligible.)
* Having undergone blood transfusion and/or a surgical procedure considered to promote anemia (excluding shunt reconstruction surgery for access to the blood) within 4 weeks before the screening assessment
* Having undergone a kidney transplantation
* Having a previous history of treatment with ASP1517.
* History of serious drug allergy including anaphylactic shock
* Participation in another clinical study or post-marketing clinical study (including that of a medical device) within 12 weeks before informed consent acquisition

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Hemoglobin (Hb) Response rate | Up to Week 24
  Hb response is defined as reaching target values for Hb and change of Hb from baseline

SECONDARY OUTCOMES:
Average Hb level from Week 18 to 24 | Week 18 to 24
Change from baseline in the average Hb level from Week 18 to 24 | Baseline and Weeks 18 to 24
Proportion of participants with the target Hb level from Week 18 to 24 | Week 18 to 24
Rate of rise in Hb levels (g/dL/week) from week 0 to at the earliest date of week 4, time of discontinuation, or time of dose adjustment | Up to Week 4
Proportion of measurement points with the target Hb level | Up to Week 24
Proportion of participants with the target Hb level at each week | Up to Week 24
Proportion of participants with the lower limit of the target Hb level | Up to Week 24
Time to achieve the lower limit of the target Hb level | Up to Week 24
Change from baseline in Hb levels to each week | Baseline and Up to Week 24
Average hematocrit level | Up to Week 24
Average reticulocyte level | Up to Week 24
Average iron (Fe) level | Up to Week 24
Average ferritin level | Up to Week 24
Average transferrin level | Up to Week 24
Average total iron binding capacity level | Up to Week 24
Average soluble transferrin receptor level | Up to Week 24
Average transferrin saturation level | Up to Week 24
Average reticulocyte hemoglobin content level | Up to Week 24
Quality of life assessed by EQ-5D-5L | Up to Week 24
  EQ-5D-5L: EuroQol 5 Dimension 5 Levels
Quality of life assessed by FACT-An | Up to Week 24
  FACT-An: Functional Assessment of Cancer Therapy-Anemia
Number of hospitalizations | Up to Week 24
Duration of hospitalizations | Up to Week 24
Safety assessed by incidence of adverse events | Up to Week 24
Number of participants with abnormal Laboratory values and/or adverse events related to treatment | Up to Week 24
Number of participants with abnormal Vital signs and/or adverse events related to treatment | Up to Week 24
Safety assessed by standard 12-lead electrocardiogram | Up to Week 24
Plasma concentration of unchanged ASP1517 | Up to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (47):
- Japan (47):
  - Site JP00003, Aichi
  - Site JP00005, Aichi
  - Site JP00042, Aichi
  - Site JP00044, Aichi
  - Site JP00020, Chiba
  - Site JP00010, Ehime
  - Site JP00021, Ehime
  - Site JP00013, Fukuoka
  - Site JP00011, Fukushima
  - Site JP00035, Fukushima
  - Site JP00017, Gifu
  - Site JP00033, Gifu
  - Site JP00012, Gunma
  - Site JP00016, Gunma
  - Site JP00025, Gunma
  - Site JP00046, Hiroshima
  - Site JP00015, Hokkaido
  - Site JP00023, Hokkaido
  - Site JP00028, Hokkaido
  - Site JP00038, Hokkaido
  - Site JP00040, Hokkaido
  - Site JP00045, Hokkaido
  - Site JP00034, Hyōgo
  - Site JP00008, Ibaraki
  - Site JP00018, Ibaraki
  - Site JP00027, Ibaraki
  - Site JP00030, Ibaraki
  - Site JP00022, Ishikawa
  - Site JP00041, Kagoshima
  - Site JP00031, Kumamoto
  - Site JP00037, Kumamoto
  - Site JP00009, Nagano
  - Site JP00014, Nagano
  - Site JP00026, Nagano
  - Site JP00047, Nagano
  - Site JP00002, Niigata
  - Site JP00029, Niigata
  - Site JP00039, Okayama
  - Site JP00024, Okinawa
  - Site JP00036, Osaka
  - Site JP00006, Saitama
  - Site JP00032, Shizuoka
  - Site JP00043, Tokushima
  - Site JP00048, Tokyo
  - Site JP00007, Tottori
  - Site JP00019, Toyama
  - Site JP00004, Yamaguchi

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Hamano T, Yamaguchi Y, Goto K, Mizokawa S, Ito Y, Dellanna F, Barratt J, Akizawa T. Risk Factors for Thromboembolic Events in Patients With Dialysis-Dependent CKD: Pooled Analysis of Phase 3 Roxadustat Trials in Japan. Adv Ther. 2024 Apr;41(4):1526-1552. doi: 10.1007/s12325-023-02727-3. Epub 2024 Feb 16. PMID 38363463
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=357